CLINICAL TRIAL: NCT03433638
Title: Retrospective Descriptive Study of Juvenile Dermatomyositis in Alsace
Brief Title: Juvenile Dermatomyositis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6785
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Juvenile Dermatomyositis
Keywords: Juvenile dermatomyositis; Inflammatory myopathy; Clinical features; Treatment
MeSH Terms: conditions — Dermatomyositis; Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective descriptive cross-sectional and observational multicenter clinical and progressive study of juvenile dermatomyositis. The aim is to determine the clinical, paraclinical, and evolutive characteristics and therapeutic modalities from a series of juvenile dermatomyositis identified in Alsace between 2000 to 2015.

ELIGIBILITY:
Inclusion Criteria:

* Age under 16 years
* Have a dermatomyositis according to the diagnostic criteria of Bohan and Peter of 1975

Exclusion Criteria:

* Refusal to participate in the study

Ages: 1 Day to 16 Years | Sex: All
Age Groups: Child
Study Population: Patient who have a dermatomyositis according to the diagnostic criteria of Bohan and Peter of 1975
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Study of clinical characteristics of juvenile dermatomyositis | The period from from January 1st, 2000 to December 31st, 2015 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Dermatologie, Strasbourg, France